CLINICAL TRIAL: NCT02959190
Title: A Phase 3, Long-Term, Open-Label Safety Study of LY2951742 (Galcanezumab) in Japanese Patients With Migraine
Brief Title: A Study of LY2951742 (Galcanezumab) in Japanese Participants With Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16108; I5Q-JE-CGAP (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-11-07; First posted 2016-11-08 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2019-08

CONDITIONS: Migraine
Keywords: prevention; prophylaxis; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — galcanezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- 120mg/120mg Galcanezumab - Episodic Migraine (EM) (Experimental): 240 milligram (loading dose) of Galcanezumab at first dosing visit followed by 120 milligram (mg) once a month for a year by subcutaneous (SC) injection. EM participants (pts) rolled over from CGAN (NCT02959177) 120 mg Galcanezumab.
  Interventions: Drug: Galcanezumab
- 240mg/240mg Galcanezumab - EM (Experimental): 240 mg Galcanezumab given SC once a month for a year. EM participants rolled over from CGAN (NCT02959177) 240 mg Galcanezumab.
  Interventions: Drug: Galcanezumab
- Placebo/ 120mg Galcanezumab - EM (Experimental): 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by SC injection. EM participants rolled over from CGAN (NCT02959177) placebo.
  Interventions: Drug: Galcanezumab
- Placebo/ 240mg Galcanezumab - EM (Experimental): 240 mg Galcanezumab given SC once a month for a year. EM participants rolled over from CGAN (NCT02959177) Placebo.
  Interventions: Drug: Galcanezumab
- 120mg Galcanezumab - CM (Experimental): 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by SC injection. Participants with CM were enrolled.
  Interventions: Drug: Galcanezumab
- 240mg Galcanezumab - CM (Experimental): 240 mg Galcanezumab given SC once a month for a year. Participants with CM were enrolled.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of the study drug known as Galcanezumab in Japanese participants with migraine.

ELIGIBILITY:
Inclusion Criteria:

* For Episodic Migraine participants: Participants who completed the treatment period of Galcanezumab study CGAN.
* Have a diagnosis of chronic migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines (1.3) (ICHD-3 2013), with a history of migraine headaches of at least 1 year prior to screening, and migraine onset prior to age 50.

Exclusion Criteria:

* For Chronic Migraine participants:

  * Are currently enrolled in or have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product.
  * Current use or prior exposure to Galcanezumab or other antibodies of calcitonin gene-related peptide (CGRP) or its receptor.
  * Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to Galcanezumab and the excipients in the investigational product.
  * History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine) defined by IHS ICHD-3 beta.
  * Failure to respond to 3 or more adequately dosed migraine preventive treatments from different classes (that is, maximum tolerated dose for at least 2 months).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- Japan (37):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chofu-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Higashiosaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iruma-Gun
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaisho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanoya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kasaoka-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kasuga-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minatoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morioka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Narashino-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nishinomiya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ota-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ōsaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōta-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saijo-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shibuya-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tachikawa-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and european union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Takeshima T, Doi H, Ooba S, Tanji Y, Ozeki A, Komori M. Clinical Evaluation After Discontinuation of Galcanezumab in Japanese Patients with Episodic and Chronic Migraine: Analysis of a Randomized, Placebo-Controlled Trial and Open-label Extension Study. Neurol Ther. 2024 Jun;13(3):697-714. doi: 10.1007/s40120-024-00602-z. Epub 2024 Apr 6. PMID 38581615
- [Derived] Hirata K, Takeshima T, Sakai F, Tatsuoka Y, Suzuki N, Igarashi H, Nakamura T, Ozeki A, Yamazaki H, Skljarevski V. A long-term open-label safety study of galcanezumab in Japanese patients with migraine. Expert Opin Drug Saf. 2021 Jun;20(6):721-733. doi: 10.1080/14740338.2021.1866536. Epub 2021 Jan 4. PMID 33393835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Episodic migraine (EM) participants rolled over from parental Study I5Q-JE-CGAN (CGAN - NCT02959177)), and chronic migraine (CM) participants were newly enrolled in this CGAP study.
Groups:
- 120 mg Galcanezumab EM: 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by subcutaneous (SC) injection. EM participants (pts) rolled over from CGAN (NCT02959177) 120 mg Galcanezumab or placebo. Participants did not receive any intervention during post-treatment follow-up phase.
- 240 mg Galcanezumab EM: 240 mg Galcanezumab given SC once a month for a year. EM participants rolled over from CGAN (NCT02959177) 240 mg Galcanezumab or placebo. Participants did not receive any intervention during post-treatment follow-up phase.
- 120 mg Galcanezumab CM: 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by SC injection. Participants with CM were enrolled. Participants did not receive any intervention during post-treatment follow-up phase.
- 240 mg Galcanezumab CM: 240 mg Galcanezumab given SC once a month for a year. Participants with CM were enrolled. Participants did not receive any intervention during post-treatment follow-up phase.
Period: Open Label
Arm/Group | 120 mg Galcanezumab EM | 240 mg Galcanezumab EM | 120 mg Galcanezumab CM | 240 mg Galcanezumab CM
Started | 120 | 126 | 32 | 33
Received at Least 1 Dose of Study Drug | 120 | 126 | 32 | 33
120mg/120mg Galcanezumab - EM | 58 | 0 | 0 | 0
240mg/240mg Galcanezumab - EM | 0 | 62 | 0 | 0
Placebo/ 120mg Galcanezumab - EM | 62 | 0 | 0 | 0
Placebo/ 240mg Galcanezumab - EM | 0 | 64 | 0 | 0
Completed | 113 | 110 | 28 | 27
Not Completed | 7 | 16 | 4 | 6
Not completed — Adverse Event | 5 | 7 | 3 | 4
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Period: Post Treatment Follow Up
Arm/Group | 120 mg Galcanezumab EM | 240 mg Galcanezumab EM | 120 mg Galcanezumab CM | 240 mg Galcanezumab CM
Started | 117 (Participants who discontinued open-label treatment phase had an option to enter post treatment phase) | 120 (Participants who discontinued open-label treatment phase had an option to enter post treatment phase) | 32 (Participants who discontinued open-label treatment phase had an option to enter post treatment phase) | 32 (Participants who discontinued open-label treatment phase had an option to enter post treatment phase)
Completed | 114 | 119 | 31 | 32
Not Completed | 3 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received at least 1 dose of the study drug.
Groups:
- 120mg/120mg Galcanezumab - EM: 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by SC injection. EM participants (pts) rolled over from CGAN (NCT02959177) 120 mg Galcanezumab.
- Total: Total of all reporting groups
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM | Total
Number analyzed (Participants) | 58 | 62 | 62 | 64 | 32 | 33 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.95 (10.04) | 45.47 (9.79) | 45.35 (10.69) | 45.08 (8.88) | 41.88 (9.40) | 43.70 (11.53) | 44.71 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 51 | 58 | 32 | 27 | 268
  Male | 10 | 10 | 11 | 6 | 0 | 6 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 58 | 62 | 62 | 64 | 32 | 33 | 311
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 58 | 62 | 62 | 64 | 32 | 33 | 311
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 58 | 62 | 62 | 64 | 32 | 33 | 311

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE started on or after the date and time of the first dose of study drug administered in this study, or started prior to the study drug administration but worsened after the study drug started. Clinically significant events were defined as SAEs and other non-serious adverse events (AEs). A summary of SAEs and other non-serious AEs is located in the Reported Adverse Events module.
Time Frame: Up To 16 Months
Population: All participants who were randomized and received at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 58 | 62 | 62 | 64 | 32 | 33
participants
  Any TEAE | 54 | 56 | 54 | 61 | 31 | 29
  Any SAE | 2 | 0 | 2 | 2 | 1 | 2

2. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Description: Serum Concentration of Galcanezumab at month 12 is reported.
Time Frame: Month 12: Predose
Population: All participants who were randomized and received at least 1 dose of the study drug and had evaluable galcanezumab PK data.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
nanogram/milliliter (ng/mL) | 21100 (6120) | 46000 (15300) | 21000 (7290) | 42200 (12400) | 20100 (8550) | 39600 (13600)

3. Secondary Outcome: Pharmacodynamics (PD): Plasma Concentration of Total Calcitonin Gene-Related Peptide (CGRP)
Description: Plasma Concentration of total CGRP at month 12 is reported.
Time Frame: Month 12: Predose
Population: All participants who were randomized and received at least 1 dose of the study drug and had measurable CGRP concentrations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
ng/mL | 4.51 (1.26) | 5.87 (1.45) | 4.69 (1.45) | 5.59 (1.45) | 4.37 (1.40) | 5.19 (1.52)

4. Secondary Outcome: Percentage of Participants Developing Anti-Drug Antibodies (ADA)
Description: Treatment emergent ADA will be defined as any of the following:
  A negative baseline result and a positive post-baseline ADA result with a titer ≥20. This is also called treatment-induced ADA.
  A positive baseline result and a positive post-baseline ADA result with a ≥4-fold increase in titers (for example, baseline titer of 10 increasing to ≥40 post-baseline). This is called treatment-boosted ADA.
Time Frame: Month 0, 1, 2, 3, 6, 9, 12 and 16: Predose; Month 0 and 14 days Postdose
Population: All participants who were randomized and received at least 1 dose of the study drug and had evaluable immunogenicity data.
Measure: Number; unit: percentage of participants
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 58 | 62 | 62 | 64 | 32 | 33
percentage of participants | 12.07 | 9.68 | 16.13 | 10.94 | 12.50 | 18.18

5. Secondary Outcome: Mean Change From Baseline in the Number of Migraine Headache Days (MHDs)
Description: Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Migraine Headache (EM Participants): A headache, with or without aura, of ≥30 minutes duration with both of the following required features (A and B): A) At least 2 of the following headache characteristics: Unilateral location; Pulsatile quality; Moderate or severe pain intensity; Aggravation by or causing avoidance of routine physical activity; AND B) During headache at least one of the following: Nausea and/or vomiting; Photophobia and phonophobia.
  Migraine Headache (CM Participants) : A headache, with or without aura, of greater than or equal to (≥30) minutes duration which meets criteria A and B or meets criterion C: A and B criteria as described above and criteria C) The headache is believed by the participant to be migraine at onset and is relieved by a triptan or ergot derivative.
Time Frame: Baseline, Month 12
Population: All participants who were randomized and received at least 1 dose of the study drug and had baseline and at least one post baseline value.
Measure: Mean (Standard Deviation); unit: MHDs
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
MHDs | -1.82 (2.96) | -1.49 (4.11) | -4.29 (4.07) | -3.23 (5.81) | -9.44 (6.16) | -8.97 (8.06)

6. Secondary Outcome: Mean Change From Baseline in the Number of Headache Days (HDs)
Description: A headache day is calendar day on which any type of headache occurs,(including migraine headache, probable migraine headache, and non-migraine headache).
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Headache days (HDs)
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
Headache days (HDs) | -2.37 (3.62) | -1.75 (4.57) | -5.04 (4.71) | -4.00 (5.14) | -9.30 (6.83) | -9.42 (8.37)

7. Secondary Outcome: Percentage of Participants With Meeting Criteria for Reductions From Baseline Greater Than or Equal to (≥) 50% in Number of Migraine Headache Days
Description: Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred. A 50% responder in a particular month is any participant who has a ≥50% reduction from baseline in the monthly number of migraine headache attacks in a 30-day interval.
Time Frame: Month 12
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 47 | 46 | 55 | 56 | 28 | 27
Percentage of participants | 48.9 | 45.7 | 52.7 | 46.4 | 35.7 | 51.9

8. Secondary Outcome: Mean Change From Baseline in the Number of Monthly Migraine Headache Days Requiring Medication for the Acute Treatment of Migraine Headache
Description: Migraine Headache Day (MHD) with Acute Medication Use: Calendar days on which migraine or probable migraine occurs, requiring acute medication.
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: MHDs with medication use
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
MHDs with medication use | -1.40 (2.54) | -1.00 (3.59) | -3.87 (3.84) | -3.01 (5.76) | -8.36 (6.29) | -7.43 (7.89)

9. Secondary Outcome: Mean Change From Baseline in the Number of Monthly Migraine Headache Days or Headache Days Requiring Medication for the Acute Treatment of Migraine Headache or Headache
Description: Monthly Migraine Headache Days or Headache Days Requiring Medication for the Acute Treatment of Migraine Headache or Headache: Calendar days on which headache, migraine or probable migraine occurs, requiring acute medication.
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: MHDs and HDs with medication use
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
MHDs and HDs with medication use | -1.62 (3.21) | -1.17 (3.89) | -4.47 (4.81) | -3.43 (5.53) | -8.21 (6.84) | -7.48 (8.21)

10. Secondary Outcome: Change From Baseline in the Patient Global Impression of Severity (PGI-S) Score
Description: The PGI-S scale is a patient-rated instrument that measures patients own global impression of their illness severity. The patient was instructed as follows: "Considering migraine as a chronic condition, how would you rate your level of illness?" Response options were from 1 ("normal, not at all ill") to 7 ("extremely ill").
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
score on a scale | -0.29 (0.76) | -0.04 (0.76) | -0.02 (0.66) | 0.11 (0.77) | -0.07 (1.59) | -0.81 (1.14)

11. Secondary Outcome: Change From Baseline on the Migraine Disability Assessment Test (MIDAS) Total Score
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that reflect the number of days reported as missing or with reduced productivity at work or home, and the number of days of missed social events. Each item has a numeric response range from 0 to 90 days, if days are missed from work or home they are not counted as days with reduced productivity at work or home. The numeric responses are summed to produce a total score ranging from 0 to 270, in which a higher value is indicative of more disability.
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
score on a scale | -0.38 (8.99) | -0.42 (15.94) | -8.67 (17.39) | -4.60 (12.77) | -20.71 (32.66) | -15.48 (32.26)

12. Secondary Outcome: Change From Baseline on the Migraine-Specific Quality of Life Questionnaire (MSQ) Version 2.1
Description: MSQ version 2.1 is a health status instrument,with a 4-week recall period,developed to address physical & emotional limitations of specific concern to individuals with migraine.Addressing the impact of migraine on work or daily activities,relationships with family & friends,leisure time,productivity,concentration, energy,tiredness & feelings.It consists of 14 items addressing 3 domains:(1)Role Function-Restrictive (items 1-7);(2)Role Function- Preventive (items 8-11);&(3)Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6), & are reverse-recoded (value 6 to 1) before the domain scores are calculated.Total raw scores for each domain is the sum of the final item value for all of the items in that domain.After total raw score is computed for each domain & total score, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement.
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
score on a scale
  Total Score | 1.02 (8.68) | 0.38 (11.97) | 7.51 (10.58) | 4.56 (11.22) | 19.23 (12.57) | 18.31 (15.67)
  Role Function-Restrictive Domain | 1.68 (9.77) | 0.22 (13.75) | 8.77 (12.74) | 4.96 (12.60) | 22.65 (15.08) | 22.96 (17.69)
  Role Function-Preventive Domain | 0.09 (9.70) | 0.75 (13.17) | 7.16 (10.18) | 3.77 (12.86) | 15.89 (13.68) | 13.52 (16.63)
  Emotional Function Domain | 0.71 (10.54) | 0.25 (11.47) | 5.06 (11.47) | 4.68 (12.34) | 15.71 (13.96) | 13.83 (17.82)

13. Secondary Outcome: Percentage of Participants With Positive Responses on Patient Satisfaction With Medication Questionnaire-Modified (PSMQ-M)
Description: The PSMQ-M is a self-rated scale which measures participants level of satisfaction with study medication.The scale has been modified for use in this study, assessing 3 items related to the clinical trial treatment over the past 4 weeks: satisfaction, preference, and side effects.Satisfaction responses range from "very unsatisfied" to "very satisfied" with the current treatment (5 categories). Preference compared the current study medication to previous medications, with responses from "much rather prefer my previous medication" to "much rather prefer the medication administered to me during the study" (5 categories). The side effects responses range from "significantly less side effects" to "significantly more side effects" (5 categories). Positive responses for each item were defined as follows: Satisfaction: "Very Satisfied" or "Somewhat Satisfied"; Preference: "Much Prefer Study Medication" or "Prefer Study Medication"; Side Effects: "Much-Less Side Effects" or "Less Side Effects".
Time Frame: Month 12
Population: All participants who were randomized and received at least 1 dose of the study drug and had month 12 PSMQ-M measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | 120mg/120mg Galcanezumab - EM | 240mg/240mg Galcanezumab - EM | Placebo/ 120mg Galcanezumab - EM | Placebo/ 240mg Galcanezumab - EM | 120mg Galcanezumab - CM | 240mg Galcanezumab - CM
Number analyzed (Participants) | 56 | 53 | 58 | 57 | 28 | 27
Percentage of participants
  Responder for satisfaction | 80.4 | 73.6 | 72.4 | 73.7 | 82.1 | 74.1
  Responder for preference | 76.8 | 73.6 | 75.9 | 75.4 | 85.7 | 81.5
  Responder for side effect | 78.6 | 69.8 | 72.4 | 71.9 | 82.1 | 81.5

ADVERSE EVENTS:
Time Frame: Up To 16 Months
Description: All participants who were randomized and received at least 1 dose of the study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- 120mg/120mg Galcanezumab - Open-Label Treatment Phase (Ph) -EM: 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by SC injection. EM participants (pts) rolled over from CGAN (NCT02959177) 120 mg Galcanezumab.
- 240mg/240mg Galcanezumab - Open-Label Treatment Ph-EM: 240 mg Galcanezumab given SC once a month for a year. EM participants rolled over from CGAN (NCT02959177) 240 mg Galcanezumab.
- Placebo/ 120mg Galcanezumab - Open-Label Treatment - EM: 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by SC injection. EM participants rolled over from CGAN (NCT02959177) placebo.
- Placebo/ 240mg Galcanezumab - Open-Label Treatment-EM: 240 mg Galcanezumab given SC once a month for a year. EM participants rolled over from CGAN (NCT02959177) Placebo.
- 120mg Galcanezumab - Open-Label Treatment Phase-CM: 240 mg (loading dose) of Galcanezumab at first dosing visit followed by 120 mg once a month for a year by SC injection. Participants with CM were enrolled.
- 240mg Galcanezumab - Open-Label Treatment Phase-CM: 240 mg Galcanezumab given SC once a month for a year. Participants with CM were enrolled.
- 120mg Galcanezumab - Post-Treatment Phase - EM; 240mg Galcanezumab - Post-Treatment Phase - EM; 120mg Galcanezumab - Post-Treatment Phase - CM; 240mg Galcanezumab - Post-Treatment Phase - CM: Participants didn't received any intervention
Arm/Group | 120mg/120mg Galcanezumab - Open-Label Treatment Phase (Ph) -EM | 240mg/240mg Galcanezumab - Open-Label Treatment Ph-EM | Placebo/ 120mg Galcanezumab - Open-Label Treatment - EM | Placebo/ 240mg Galcanezumab - Open-Label Treatment-EM | 120mg Galcanezumab - Open-Label Treatment Phase-CM | 240mg Galcanezumab - Open-Label Treatment Phase-CM | 120mg Galcanezumab - Post-Treatment Phase - EM | 240mg Galcanezumab - Post-Treatment Phase - EM | 120mg Galcanezumab - Post-Treatment Phase - CM | 240mg Galcanezumab - Post-Treatment Phase - CM
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/62 | 0/62 | 0/64 | 0/32 | 0/33 | 0/117 | 0/120 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/58 | 0/62 | 2/62 | 2/64 | 1/32 | 2/33 | 2/117 | 1/120 | 1/32 | 1/32
Other Adverse Events (participants affected / at risk) | 54/58 | 56/62 | 54/62 | 61/64 | 31/32 | 29/33 | 40/117 | 37/120 | 10/32 | 13/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 120mg/120mg Galcanezumab - Open-Label Treatment Phase (Ph) -EM (N=58) | 240mg/240mg Galcanezumab - Open-Label Treatment Ph-EM (N=62) | Placebo/ 120mg Galcanezumab - Open-Label Treatment - EM (N=62) | Placebo/ 240mg Galcanezumab - Open-Label Treatment-EM (N=64) | 120mg Galcanezumab - Open-Label Treatment Phase-CM (N=32) | 240mg Galcanezumab - Open-Label Treatment Phase-CM (N=33) | 120mg Galcanezumab - Post-Treatment Phase - EM (N=117) | 240mg Galcanezumab - Post-Treatment Phase - EM (N=120) | 120mg Galcanezumab - Post-Treatment Phase - CM (N=32) | 240mg Galcanezumab - Post-Treatment Phase - CM (N=32)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0/48 (0) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 1/105 (1) | 0 (0) | 0/26 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1/48 (1) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 120mg/120mg Galcanezumab - Open-Label Treatment Phase (Ph) -EM (N=58) | 240mg/240mg Galcanezumab - Open-Label Treatment Ph-EM (N=62) | Placebo/ 120mg Galcanezumab - Open-Label Treatment - EM (N=62) | Placebo/ 240mg Galcanezumab - Open-Label Treatment-EM (N=64) | 120mg Galcanezumab - Open-Label Treatment Phase-CM (N=32) | 240mg Galcanezumab - Open-Label Treatment Phase-CM (N=33) | 120mg Galcanezumab - Post-Treatment Phase - EM (N=117) | 240mg Galcanezumab - Post-Treatment Phase - EM (N=120) | 120mg Galcanezumab - Post-Treatment Phase - CM (N=32) | 240mg Galcanezumab - Post-Treatment Phase - CM (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness transitory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cyst (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 3 (3) | 3 (3) | 7 (7) | 5 (5) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oesophageal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (4) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site eczema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 11 (37) | 15 (66) | 11 (53) | 16 (50) | 3 (4) | 3 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 3 (3) | 2 (3) | 2 (6) | 7 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (2) | 3 (7) | 4 (5) | 11 (31) | 2 (2) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 7 (26) | 9 (22) | 10 (33) | 17 (68) | 5 (9) | 4 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (13) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 6 (17) | 5 (12) | 4 (12) | 7 (17) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoviral conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 4 (6) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 5 (6) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 11 (11) | 8 (8) | 5 (5) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 27 (44) | 29 (45) | 25 (44) | 32 (48) | 13 (19) | 16 (23) | 9 (10) | 8 (8) | 2 (2) | 2 (3)
Oral herpes (Infections and infestations) | 2 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0/48 (0) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 1/105 (1) | 0 (0) | 0/26 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1/48 (1) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Viral tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/48 (0) | 1/52 (1) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 1/96 (1) | 0/105 (0) | 0 (0) | 0/26 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anti-cyclic citrullinated peptide antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/48 (2) | 0/52 (0) | 0/51 (0) | 1/58 (1) | 1 (1) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thunderclap headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/48 (0) | 0/52 (0) | 0/51 (0) | 1/58 (1) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frustration tolerance decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1/48 (1) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1/48 (1) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Cervical polyp (Reproductive system and breast disorders) | 0/48 (0) | 0/52 (0) | 0/51 (0) | 1/58 (1) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/48 (1) | 1/52 (1) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 1/96 (1) | 1/105 (1) | 0 (0) | 0/26 (0)
Endometriosis (Reproductive system and breast disorders) | 1/48 (1) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Menopausal disorder (Reproductive system and breast disorders) | 0/48 (0) | 1/52 (1) | 0/51 (0) | 1/58 (1) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1/48 (1) | 0/52 (0) | 0/51 (0) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 1/105 (1) | 0 (0) | 0/26 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/48 (0) | 0/52 (0) | 1/51 (1) | 0/58 (0) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/48 (0) | 0/52 (0) | 0/51 (0) | 1/58 (1) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1/48 (1) | 1/52 (1) | 0/51 (0) | 2/58 (3) | 0 (0) | 0/27 (0) | 0/96 (0) | 1/105 (1) | 1 (1) | 0/26 (0)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (5) | 4 (4) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria thermal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone graft (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical polypectomy (Surgical and medical procedures) | 0/48 (0) | 0/52 (0) | 0/51 (0) | 1/58 (1) | 0 (0) | 0/27 (0) | 0/96 (0) | 0/105 (0) | 0 (0) | 0/26 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin cyst excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon sheath incision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review the study result with PIs prior to public release and can embargo a communication about it until the public release by the contract with Investigator sites.

DOCUMENTS (3):
  • Study Protocol: CGAP Protocol (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02959190/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02959190/SAP_001.pdf
  • Study Protocol: CGAP (1) Protocol Addendum (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02959190/Prot_002.pdf